CLINICAL TRIAL: NCT03481192
Title: Voluntary Drug Poisoning by Psychoactive Molecules: Identify Cognitive Markers Predictive of a Preserved Memory of Care in Psychiatric Emergencies
Brief Title: Voluntary Drug Poisoning by Psychoactive Molecules: Identify Cognitive Markers
Acronym: IMG-COG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/17/0160; 2017-A01581-52 (Other: ID-RCB)
Record Dates: First submitted 2018-03-07; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Suicide; Drug Poisoning
MeSH Terms: conditions — Suicide; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: To groups of patients :
  A group of patients admitted for IMV exclusively using amnesic substances.
  A control group admitted for IMV and ingested exclusively non-amnesic
  Two visits, the first one for the first evaluation of cognitive functions directly following the psychiatric interview (E1), and the second one at 24h-48h after the psychiatric evaluation (E2)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group using amnesic substances (Experimental): A group of patients admitted for IMV exclusively using amnesic substances. Benzodiazepines, benzodiazepines, tricyclic antidepressants, neuroleptics, antihistamines, other atropine substances, anti-epileptics and opiates.
  Two visits for evaluation, the first one for the first evaluation of cognitive functions directly following the psychiatric interview, and the second one at 24h-48h of the psychiatric evaluation (T2), a second evaluation (E2) will take place.
  Interventions: Behavioral: Two visits for evaluation
- A control group (Active Comparator): A control group that ingested exclusively non-amnesic substances among them most frequently ingested in this context, ie the following classes: level 1 analgesics, antibiotics, serotonergic and noradrenergic antidepressants, oral antidiabetic, thyroid hormones, anti oral coagulant.
  Two visits for evaluation, the first one for the first evaluation of cognitive functions directly following the psychiatric interview, and the second one at 24h-48h of the psychiatric evaluation (T2), a second evaluation (E2) will take place.
  Interventions: Behavioral: Two visits for evaluation

INTERVENTIONS:
Behavioral: Two visits for evaluation — Visit 1:The first evaluation (E1) of cognitive functions will take place directly following the psychiatric interview (T1), in order to better reflect the cognitive abilities at the time of the proposal of the care project.
  This will include the Memory Functioning Questionnaire (MFQ), the five words of DUBOIS, the TMT-A and B, the WAIS code test, and the BADDELEY door test. An intercurrent type ringing event of the phone will take place during this evaluation.
  Visit 2: At 24h-48h of the psychiatric evaluation (T2), a second evaluation (E2) will take place.
  An episodic memory score will be determined by asking the patient to recall,as precisely as possible the evaluation E1. At first the reminder will be free,the data can be completed, if necessary, with an indication, a recognition.

SUMMARY:
To identify in patients admitted for Voluntary drug poisoning (IMV) by psychoactive substances, T1 predictors of T2 recall of psychiatric interview and care project.

DETAILED DESCRIPTION:
The methodology will compare the episodic memory results of patients admitted for IMV who have exclusively ingested amnesic substances to a subject control group that has made IMV with non-amnesic substances such as paracetamol. The purpose of this comparison is to ensure that memory problems are not related to the context of the suicidal crisis.

The second step will be able to relate the memory score of the predictor variables. To achieve this, it will perform a multivariate linear regression in each group in order to confirm the results of the pilot study and to be able to regress in the control group which was not possible in the pilot study because of the lack of effective.

Finally, this study will try to establish, using Receiver Operating Characteristic (ROC) curves, thresholds for cognitive scores and begin to develop a tool for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Group amnesic substances :

* Age from 18 to 65 years
* Admitted to emergencies for IMV by benzodiazepines
* Supported at Toulouse University Hospital (hospitalization, outpatient)

Group control :

* Age from 18 to 65 years
* Admitted to emergencies for IMV by non-depressive substances of the central nervous system
* Supported at Toulouse University Hospital (hospitalization, outpatient)

Exclusion Criteria:

* Cognitive Disorder Due to an Organic Disorder Neuro Degenerative Disease, Korsakoff Syndrome) or Mental Retardation Diagnosed
* Patient under guardianship
* Not speaking and / or not reading French
* Neurodegenerative disease diagnosed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the episodic score recall of the first interview (T1) at T2 | Just After/24-48h after the psychiatric interview
  This score is based on the episodic scale. The episodic score is a reflection of the patient's memory of the emergency psychiatric assessment. In this study, this score will be used as a variable independent of the multivariate linear regression, the objective of the study being to identify the variables significantly related to this score.
  The total episodicity score is calculated by adding the episodic scores of several events. A continuous score is obtained and between 0 and 38.

SECONDARY OUTCOMES:
Comparison of cognitive scores between the amnesic substances group and the control group using the The Memory Functioning Questionnaire (MFQ) abridged version of tthe Memory Functioning Questionnaire | Just After/24-48h after the psychiatric interview
  The control group is a group of subject having made an IMV with non-amnesic substances such as paracetamol.
Sensitivity score of each test for the episodic memory test | Just After/24-48h after the psychiatric interview
  Sensitivity score of each test
Specificity score of each test for the episodic memory test | Just After/24-48h after the psychiatric interview
  Specificity score of each test

CONTACTS AND LOCATIONS:
Overall Officials: Juliette SALLES, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No